CLINICAL TRIAL: NCT03204188
Title: A Phase II Study Of Ibrutinib, Fludarabine, and Pembrolizumab in High-Risk or Relapsed/Refractory Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (CLL/SLL)
Brief Title: Ibrutinib, Fludarabine, and Pembrolizumab in High-Risk or Relapsed/Refractory Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 170118; 17-H-0118
Record Dates: First submitted 2017-06-28; First posted 2017-06-29 (Actual); Results first posted 2023-04-19 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: B-Cell Chronic Lymphocytic Leukemia; B-Lymphocytic Leukemia, Chronic; Chronic Lymphocytic Leukemia; Leukemia, Chronic Lymphatic; Leukemia, Chronic Lymphocytic, B-Cell; Leukemia, Lymphocytic, Chronic; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphocytic Leukemia, Chronic, B Cell; Lymphocytic Leukemia, Chronic, B-Cell
Keywords: Deletion 17p; TP53 Mutation; NOTCH1 mutation; Complex Cytogenetics; Bruton's Tyrosine Kinase (BTK) Inhibitor
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Chromosome 17 deletion | interventions — ibrutinib; fludarabine; fludarabine phosphate; pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ibrutinib, Fludarabine, and Pembrolizumab in Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (Experimental): Ibrutinib, Fludarabine, and Pembrolizumab combination therapy will be administered in participants with High-Risk or Relapsed/Refractory Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (CLL/SLL). Ibrutinib will be administered daily by mouth starting cycle -3 at 420 mg until end study or disease progression or intolerable side effects occur. Fludarabine will be administered intravenously only on cycle -2 at 25mg/m^2 x5 days. Pembrolizumab will be administered intravenously every 3 weeks at 200 mg starting from cycle 1 through cycle 17 or 1 year of immunotherapy phase.
  Interventions: Drug: Ibrutinib; Drug: Fludarabine; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Ibrutinib — Ibrutinib will be administered daily by mouth starting cycle -3 at 420 mg until end study or disease progression or intolerable side effects occur.
  Other Names: Imbruvica
Drug: Fludarabine — Fludarabine will be administered intravenously only on cycle -2 at 25mg/m^2 x5 days.
  Other Names: Fludara
Drug: Pembrolizumab — Pembrolizumab will be administered intravenously every 3 weeks at 200 mg starting from cycle 1 through cycle 17 or 1 year of immunotherapy phase.
  Other Names: Keytruda

SUMMARY:
Background:

Chronic lymphocytic leukemia and small lymphocytic lymphoma (hereby referred as CLL) are tumors of B cells. A subset of patients categorized as high-risk CLL has a poor clinical outcome when treated with conventional chemotherapy. This single-arm, phase II study investigates the combination of ibrutinib, fludarabine and pembrolizumab for treatment of CLL. Ibrutinib is an orally administered therapy for CLL. Fludarabine is a well-tolerated drug that has been widely used to treat CLL. Also, fludarabine can modulate CLL cells as well as immune cells that support the growth of CLL cells. Pembrolizumab recruits immune cells to attack CLL cells. With this approach we hope to achieve a greater reduction in CLL cells than with single agent ibrutinib and to restore healthier immune system that could contribute to durable responses.

Objective:

To investigate the rate of complete response to ibrutinib, short course fludarabine and pembrolizumab.

Eligibility:

Patients with active CLL meeting treatment indications defined by 2008 International Workshop on CLL (IWCLL) consensus guideline.

High-risk CLL defined by one of the following:

* Relapsed/refractory disease status, or
* Presence of high-risk mutations regardless of prior treatment status: deletion 17p, TP53 mutation, NOTCH1 mutation, SF3B1 mutation, MYC aberration, or complex cytogenetics.

Design:

This is a single-arm, open-label phase II study.

Timeline: Treatment on this study is given in cycles from cycle -3 to 17, then in months beyond cycle 17. Cycles -3 to -1 are 28-day cycles. Cycles 1 to 17 are 21-day cycles. After completion of 1 year of pembrolizumab, the time on study is by chronological months on study from starting pembrolizumab.

Treatment plan:

* Ibrutinib is given starting from cycle -3 and continuously until disease progression or intolerable side effects occur.
* Fludarabine is given on D1-D5 on cycle -2 only
* Pembrolizumab is given every 3 weeks starting from cycle 1 for 1 year.
* Minimal residual disease will be measured at 2 years from cycle 1 to determine the need for long- term treatment with ibrutinib.

  * Previously-untreated patients who achieve minimal residual disease negativity will stop ibrutinib.
  * Patients who do not achieve minimal residual disease negativity or who has Relapsed/refractory CLL will continue ibrutinib.

DETAILED DESCRIPTION:
Background:

This study investigates the combination of ibrutinib, fludarabine and pembrolizumab for treatment of CLL. Chronic lymphocytic leukemia and small lymphocytic lymphoma (hereby referred as CLL) are tumors of B cells. A subset of patients categorized as high-risk CLL has a poor clinical outcome when treated with conventional chemotherapy. High-risk CLL is defined by relapsed/refractory disease status, or the presence of high-risk mutations, such as deletion 17p, TP53, and NOTCH1. While the cause of CLL is still unclear, studies have indicated critical factors required for the tumor cells. First, CLL cells grow and survive because they receive signals through the B-cell receptor (BCR); and second, CLL cells benefit from interactions with other cells, especially T cells.

The stimulation through the BCR can be blocked by ibrutinib, which is an oral drug that selectively inhibits Bruton's tyrosine kinase (BTK). In clinical trials, ibrutinib demonstrated safety and high response rates in patients with high-risk disease. Ibrutinib has gained FDA approval as a treatment for CLL regardless of prior treatment or cytogenetic status. However, single-agent ibrutinib has limitations; the drug does not eliminate all tumor cells and, with time, the tumor cells may become resistant. Therefore, combination of ibrutinib with other drugs could be beneficial.

Objectives:

-To investigate the rate of complete response to ibrutinib, short course fludarabine and pembrolizumab.

Key eligibility criteria:

Patients with active CLL meeting treatment indications defined by 2008 International Workshop on CLL (IWCLL) consensus guideline.

High-risk CLL defined by one of the following:

Relapsed/refractory disease status, or

Presence of high-risk mutations regardless of prior treatment status: deletion 17p, TP53 mutation, NOTCH1 mutation, SF3B1 mutation, MYC aberration, or complex cytogenetics.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Men and women with histologically confirmed CLL or SLL
* Active disease as defined by at least one of the following IWCLL consensus criteria:

  * Weight loss greater than or equal to 10% within the previous 6 months.
  * Extreme fatigue.
  * Fevers of greater than 100.5 degrees F for greater than or equal to 2 weeks without evidence of infection.
  * Night sweats for more than one month without evidence of infection.
  * Evidence of progressive marrow failure as manifested by the development of, or worsening of, anemia and/or thrombocytopenia.
  * Massive or progressive splenomegaly.
  * Massive nodes or clusters or progressive lymphadenopathy.
  * Progressive lymphocytosis with an increase of >50% over a 2-month period, or an anticipated doubling time of less than 6 months.
* High-risk disease defined by meeting at least one of the following three criteria:

  * Relapsed and/or refractory CLL/SLL.
  * Presence of high-risk mutations detected by FISH or targeted sequencing, regardless of prior treatments status.

    * FISH: deletion 17p (or TP53), complex cytogenetics (3 or more abnormalities)
    * Targeted sequencing: TP53 mutations, SF3B1 mutations, or NOTCH1 mutation. Pathologic mutations occurring at the coding regions are accepted as relevant mutations.
    * MYC aberration. Aberration includes rearrangement, amplification, and tissue expression by immunohistochemistry
  * CLL or SLL with disease transformation with Hodgkin-like cells regardless of prior treatment status.
* Eastern Cooperative Oncology Group (ECOG) performance status of less than or equal to 1.
* Adequate organ function as defined by the study protocol.
* Agreement to use acceptable methods of contraception during the study and for 90 days after the last dose of study drug if sexually active and able to bear or beget children.
* Willing and able to participate in all required evaluations and procedures in this study protocol including swallowing capsules without difficulty.
* Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information.
* Individuals greater than or equal to 18 years old

EXCLUSION CRITERIA:

* Transformation of CLL into lymphomas other than those with Hodgkin-like cells.
* Currently receiving or previously participated to receive an investigational agent within 4 weeks prior to study treatment.
* Currently receiving or previously received monoclonal antibodies, immunomodulatory therapy, chemotherapy, radiation, or radioimmunotherapy within 4 weeks prior to study treatment, or has not recovered from non-hematologic adverse events due to a previously administered agent.
* Major surgery within 4 weeks of first dose of study drug
* Currently receiving systemic steroid therapy (i.e. prednisone) or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Prior therapy with BTK inhibitor, anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
* Active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g.., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Known additional malignancy that is progressing or requires active treatment.
* Known history of, or any evidence of active, non-infectious pneumonitis that required steroids.
* Known bleeding disorders (i.e., von Willebrand s disease or hemophilia).
* Known HIV infection
* Active hepatitis B or hepatitis C infection.
* Recent known active infection requiring systemic therapy that was completed less than or equal to 14 days before the first dose of study drug.
* Known history of active tuberculosis.
* Any uncontrolled active systemic infection.
* Known hypersensitivity to ibrutinib, fludarabine, or pembrolizumab.
* Requires concomitant anticoagulation with Coumadin (warfarin) or other vitamin K antagonists.
* Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel or ulcerative colitis, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction
* History of stroke or intracranial hemorrhage within 6 months before the first dose of study drug
* Subjects who received a strong cytochrome P450 (CYP) 3A inhibitor within 7 days prior to the first dose of ibrutinib or subjects who require continuous treatment with a strong CYP3A inhibitor
* Currently active, clinically significant cardiovascular disease including uncontrolled or symptomatic arrhythmias, Class 3 or 4 congestive heart failure as defined by New York Heart Association Functional Classification, or a history of myocardial infarction, unstable angina or acute coronary syndrome within 6 months of screening.
* Life-threatening illness, medical condition or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of ibrutinib and fludarabine, or put the study outcomes at undue risk
* Female patients who are currently in pregnancy, or unwilling to use acceptable methods of contraception or refrain from pregnancy if of childbearing potential or currently breastfeeding. Male patients who are unwilling to follow the contraception requirements described in this protocol.
* Psychiatric illness/social situations that would limit the patient s ability to tolerate and/or comply with study requirements.
* Unable to understand the investigational nature of the study or give informed consent.
* Currently active, clinically significant hepatic impairment Child-Pugh class B or C according to the Child Pugh classification.
* Vaccinated with live, attenuated vaccines within 4 weeks of first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-09-22 (Actual); Primary Completion 2022-07-18 (Actual); Study Completion 2026-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adrian U Wiestner, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2017-H-0118.html

RESULTS

PARTICIPANT FLOW:
Period: Conditioning Phase (12 Weeks)
Arm/Group | Ibrutinib, Fludarabine, and Pembrolizumab in Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
Started | 15
Completed | 15
Not Completed | 0
Period: Immunotherapy Phase (1 Year)
Arm/Group | Ibrutinib, Fludarabine, and Pembrolizumab in Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
Started | 15
Completed | 10
Not Completed | 5
Not completed — Adverse Event | 4
Not completed — Death | 1
Period: Follow-up Phase (Extension Study)
Arm/Group | Ibrutinib, Fludarabine, and Pembrolizumab in Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
Started | 10
Completed | 4
Not Completed | 6
Not completed — Progression of Disease | 4
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Arm/Group | Ibrutinib, Fludarabine, and Pembrolizumab in Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 11
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Response of the Combination of Ibrutinib, Fludarabine, and Pembrolizumab in Patients With High-risk and/or Relapsed/Refractory Chronic Lymphocytic Leukemia and Small Lymphocytic Leukemia
Description: Rate of complete response with combination ibrutinib, fludarabine, and pembrolizumab in patients with high-risk and/or relapsed/refractory chronic lymphocytic leukemia and small lymphocytic leukemia. Response assessments defined by IWCLL 2008 guidelines incorporating the 2012 and 2013 clarifications for patients treated with kinase inhibitors. Complete response defined as: Lymphadenopathy is none > 1.5 cm; No Splenomegaly or Hepatomegaly; Blood Lymphocytes <4000/uL; Bone Marrow is normocellular, <30% lymphocytes, no B-lymphoid nodules; Platelet count >100,000/uL; Hemoglobin > 11.0 g/dL and Neutrophils >1500/uL. Partial response is defined by meeting 2 criteria: Lymphadenopathy decrease > or = 50%; Splenomegaly or Hepatomegaly decrease > or = 50%; Blood Lymphocytes decrease > or = 50% from baseline; Platelet is > 100,000/uL or increase > or = 50% over baseline; Hemoglobin is > 11.0 g/dL or increase > or = 50% over baseline; Neutrophils is > 1500/uL or increase > or = 50% over baseline.
Time Frame: 1 year
Population: Includes all participants that completed the 1 year evaluation
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrutinib, Fludarabine, and Pembrolizumab in Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
Number analyzed (Participants) | 10
Participants
  Complete Response | 1
  Partial Response | 9

2. Secondary Outcome: Tolerability, Response and Best Response, Survival
Description: Tolerability of the combination regimen, Overall response rate (ORR), Duration of response (DOR), Best response, Minimal residual disease (MRD) status, Progression-free survival (PFS), Overall survival (OS), To explore the biologic effects on B- and T-cell subsets and function, To identify predictors of clinical response.
Time Frame: 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 5 year
Arm/Group | Ibrutinib, Fludarabine, and Pembrolizumab in Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
All-Cause Mortality (participants affected / at risk) | 1/15
Serious Adverse Events (participants affected / at risk) | 11/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ibrutinib, Fludarabine, and Pembrolizumab in Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (N=15)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (2)
Malaise (General disorders) | 1 (1)
Multi-organ failure (General disorders) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 2 (6)
Sepsis (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Prostatic adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (4)
Kidney infection (Renal and urinary disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ibrutinib, Fludarabine, and Pembrolizumab in Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (N=15)
Anemia (Blood and lymphatic system disorders) | 7 (13)
Hepatosplenomegaly (Blood and lymphatic system disorders) | 1 (1)
Iron deficiency anemia (Blood and lymphatic system disorders) | 1 (2)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (4)
Fullness above his left collar bone (Blood and lymphatic system disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (2)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
AV nodal disease (Cardiac disorders) | 1 (1)
Abnormal R-wave progression, early transition of QRS (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1)
Non-specific T wave abnormalities (Cardiac disorders) | 1 (1)
Premature ventricular complex (PVC) (Cardiac disorders) | 1 (1)
Heart murmur (Cardiac disorders) | 1 (1)
Premature ventricular contractions (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 3 (5)
Pericardial effusion (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 3 (6)
Sinus tachycardia (Cardiac disorders) | 5 (6)
Supraventricular tachycardia (Cardiac disorders) | 2 (2)
Ventricular tachycardia (Cardiac disorders) | 3 (3)
Aural fullness in left ear (Ear and labyrinth disorders) | 1 (1)
Left ear pressure (Ear and labyrinth disorders) | 1 (1)
Ear bleeding (Ear and labyrinth disorders) | 1 (1)
Left Mastoid Effusion (Ear and labyrinth disorders) | 2 (2)
Right posterior tympanic membrane hemorrhage (Ear and labyrinth disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 2 (2)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Vestibular disorder (Ear and labyrinth disorders) | 1 (1)
Triiodothyronine decreased (Endocrine disorders) | 3 (4)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 4 (5)
Blurred vision (Eye disorders) | 5 (5)
Conjunctivitis (Eye disorders) | 3 (5)
Dry eye (Eye disorders) | 2 (2)
Bilateral posterior ocular capsule scarring (Eye disorders) | 1 (1)
Blepharitis (Eye disorders) | 1 (1)
Diplopia (Eye disorders) | 1 (1)
Dry macular degeneration bilaterally (Eye disorders) | 1 (1)
Eye hemorrhage (hyphema, subconjunctival hemorrhage and retinal hemorrhage) (Eye disorders) | 1 (1)
Injected conjunctiva (Eye disorders) | 1 (1)
Left eye stye (Eye disorders) | 1 (1)
Lower eyelid droop (Eye disorders) | 1 (1)
Retinal hemorrhage (Eye disorders) | 1 (1)
Vision impairment (glasses) (Eye disorders) | 1 (1)
Left sided subconjunctival hemorrhage (Eye disorders) | 1 (2)
Retinal detachment (Eye disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 5 (6)
Anorexia (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 3 (3)
Cheilitis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (2)
Dental caries (Gastrointestinal disorders) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 9 (15)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3 (3)
Aphthous ulcers (Gastrointestinal disorders) | 1 (1)
Esophageal spasm (Gastrointestinal disorders) | 1 (1)
Hiatal hernia (Gastrointestinal disorders) | 1 (1)
Hyperactive bowel sounds (Gastrointestinal disorders) | 1 (1)
Lower lip macular lesion (Gastrointestinal disorders) | 1 (1)
Oral ulcers (Gastrointestinal disorders) | 1 (1)
Right inguinal hernia (Gastrointestinal disorders) | 1 (1)
Hematochezia (Gastrointestinal disorders) | 1 (1)
Early satiety (Gastrointestinal disorders) | 1 (1)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (17)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 5 (9)
Chills (General disorders) | 1 (1)
Edema limbs (General disorders) | 9 (15)
Fatigue (General disorders) | 10 (11)
Fever (General disorders) | 3 (3)
Flu like symptoms (General disorders) | 8 (9)
Gait disturbance (General disorders) | 1 (1)
Cold intolerance (General disorders) | 1 (1)
Rhinorrhea (General disorders) | 1 (1)
Infusion site extravasation (General disorders) | 1 (1)
Localized edema (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Pain (General disorders) | 10 (15)
Sinus bradycardia (General disorders) | 1 (1)
Gallbladder obstruction (Hepatobiliary disorders) | 1 (1)
Gallstones (Hepatobiliary disorders) | 1 (1)
Hypocalcemia (Hepatobiliary disorders) | 1 (1)
Allergic reaction (Immune system disorders) | 2 (2)
Anorectal infection (Infections and infestations) | 1 (1)
Bronchial infection (Infections and infestations) | 1 (1)
COVID-19 infection (Infections and infestations) | 2 (2)
COVID-19 positive (Aptima SARS-CoV-2 assay) (Infections and infestations) | 1 (1)
COVID-19 positive PCR (Infections and infestations) | 1 (1)
HSV-1 positive oral ulcer (Infections and infestations) | 1 (1)
Shingles (Infections and infestations) | 2 (2)
Lung infection (Infections and infestations) | 3 (4)
Mucosal infection (Infections and infestations) | 2 (2)
Nail infection (Infections and infestations) | 2 (2)
Platelet count decreased (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 3 (4)
Soft tissue infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 3 (3)
Urinary tract infection (Infections and infestations) | 1 (1)
Weight gain (Infections and infestations) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 9 (11)
Burn (Injury, poisoning and procedural complications) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 5 (8)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Splinter in Right thumb (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 5 (27)
Alkaline phosphatase increased (Investigations) | 5 (5)
Aspartate aminotransferase increased (Investigations) | 7 (15)
Blood bilirubin increased (Investigations) | 6 (14)
CD4 lymphocytes decreased (Investigations) | 3 (3)
CPK increased (Investigations) | 2 (3)
Cardiac troponin T increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 5 (7)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1)
GGT increased (Investigations) | 1 (4)
Haptoglobin decreased (Investigations) | 1 (2)
Hyperglycemia (Investigations) | 1 (1)
Hypophosphatemia (Investigations) | 1 (1)
INR increased (Investigations) | 1 (1)
Ammonia level elevated (Investigations) | 1 (1)
Amylase decreased (Investigations) | 1 (1)
Blood lactate dehydrogenase decreased (Investigations) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 3 (5)
CRP increased (Investigations) | 2 (2)
Colonoscopy (Investigations) | 1 (1)
Creatine kinase decreased (Investigations) | 2 (2)
Creatinine decreased (Investigations) | 1 (2)
D-dimer increased (Investigations) | 1 (1)
HDL decreased (Investigations) | 1 (1)
Hyperphosphatemia (Investigations) | 1 (1)
Hypochloremia (Investigations) | 2 (4)
Hypogammaglobulinemia (Investigations) | 1 (1)
Hypouricemia (Investigations) | 1 (1)
Infarct in the left cerebellar vermis (Investigations) | 1 (1)
Interstitial markings bilateral lungs on CXR (Investigations) | 1 (1)
Iron deficiency (Investigations) | 1 (1)
Iron deficiency anemia (Investigations) | 1 (1)
Lactic acid increase (Investigations) | 1 (1)
Lipase decreased (Investigations) | 1 (1)
Neutrophil count increased (Investigations) | 8 (19)
Nodule in right thyroid gland (Investigations) | 1 (1)
Prostate Specific Antigen (PSA) elevated (Investigations) | 1 (1)
Serum Iron decreased (Investigations) | 1 (1)
TSH increased (Investigations) | 1 (1)
Urea nitrogen increased (Investigations) | 3 (3)
Urinalysis abnormal (Investigations) | 1 (1)
White Blood Cell increased (Investigations) | 2 (2)
Creatine kinase decreased (Investigations) | 1 (1)
Triiodothyronine decreased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 7 (52)
Lymphocyte count increased (Investigations) | 6 (8)
Neutrophil count decreased (Investigations) | 11 (39)
Platelet count decreased (Investigations) | 9 (44)
Weight gain (Investigations) | 12 (20)
Weight loss (Investigations) | 2 (2)
White blood cell decreased (Investigations) | 5 (20)
Alanine aminotransferase increased (Metabolism and nutrition disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 7 (16)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 4 (4)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 5 (11)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (5)
Hyperphosphatemia (Metabolism and nutrition disorders) | 2 (2)
Iron deficiency (Metabolism and nutrition disorders) | 1 (3)
Polydipsia (Metabolism and nutrition disorders) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 2 (3)
Obesity (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (22)
Arthritis (Musculoskeletal and connective tissue disorders) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Left Shin nodules (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasm (Musculoskeletal and connective tissue disorders) | 1 (1)
Polymyalgia rhematica (Musculoskeletal and connective tissue disorders) | 1 (1)
Restless leg syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Right Maxilla tenderness (Musculoskeletal and connective tissue disorders) | 1 (1)
Right Shin nodules (Musculoskeletal and connective tissue disorders) | 1 (1)
Right three proximal interphalangeal mild synovitis/tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Degenerative joint disease of neck (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (8)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3)
Angioma and melanocytic nevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Basal cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Left shoulder lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Sessile polyps (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Left maxillary mucous retention cyst or polyp (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Left neck nodule (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 1 (1)
Concentration impairment (Nervous system disorders) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 6 (8)
Headache (Nervous system disorders) | 8 (15)
Memory impairment (Nervous system disorders) | 1 (1)
Anisocoria (Nervous system disorders) | 1 (1)
Sciatic pain (Nervous system disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 3 (3)
Peripheral motor neuropathy (Nervous system disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 3 (3)
Insomnia (Psychiatric disorders) | 3 (3)
Suicidal ideation (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 3 (6)
Hematoma (Renal and urinary disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 4 (6)
Proteinuria (Renal and urinary disorders) | 3 (3)
Decreased urine output (Renal and urinary disorders) | 1 (1)
Renal lesion (Renal and urinary disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1)
Prostatic obstruction (Reproductive system and breast disorders) | 1 (1)
Testicular swelling (hydrocele) (Reproductive system and breast disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Mediastinal/ hilar adenopathy developing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Mosaic attenuation ground-glass pattern in both lungs (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary nodules (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 5 (5)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 (3)
Paronychia (Skin and subcutaneous tissue disorders) | 1 (1)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (5)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 (7)
Abrasion (Skin and subcutaneous tissue disorders) | 1 (1)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 2 (2)
Basal cell carcinoma (Skin and subcutaneous tissue disorders) | 1 (1)
Brittle nails (Skin and subcutaneous tissue disorders) | 4 (4)
Insect bite (Skin and subcutaneous tissue disorders) | 1 (1)
Laceration (Skin and subcutaneous tissue disorders) | 2 (2)
Laceration on finger (Skin and subcutaneous tissue disorders) | 1 (1)
Lesion (Skin and subcutaneous tissue disorders) | 1 (1)
Mosquito bites (Skin and subcutaneous tissue disorders) | 1 (1)
Multiple skin lesions (Skin and subcutaneous tissue disorders) | 1 (1)
Nodule (Skin and subcutaneous tissue disorders) | 1 (1)
Nodule-insect bite (Skin and subcutaneous tissue disorders) | 1 (1)
Non-healing lesion (Skin and subcutaneous tissue disorders) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 2 (2)
Palpable lesion on hand (Skin and subcutaneous tissue disorders) | 1 (1)
Skin lesions (Skin and subcutaneous tissue disorders) | 1 (1)
Facial bleeding (right ala of nose) (Skin and subcutaneous tissue disorders) | 1 (1)
Laceration (Skin and subcutaneous tissue disorders) | 1 (1)
Papule (Skin and subcutaneous tissue disorders) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 4 (4)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Skin infection (Skin and subcutaneous tissue disorders) | 2 (2)
Telangiectasia (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 8 (16)
Hypotension (Vascular disorders) | 5 (5)
Prostractic obstruction (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-20): https://cdn.clinicaltrials.gov/large-docs/88/NCT03204188/Prot_SAP_000.pdf